CLINICAL TRIAL: NCT06809309
Title: The Ventilation During In-Hospital Cardiac Arrest (VENT-IHCA) Study
Brief Title: The Ventilation During In-hospital Cardiac Arrest Study
Acronym: VENT-IHCA
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: VENT-IHCA; 1-16-02-301-24 (Registry Identifier: Internal Registry Central Denmark Region); 2022-0367531 (Registry Identifier: Internal Research Registry Aarhus University)
Record Dates: First submitted 2025-01-20; First posted 2025-02-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Arrest (CA); In-Hospital Cardiac Arrest; Heart Arrest
Keywords: prospective observational study; ventilation; manual ventilation; cardiac arrest; in-hospital cardiac arrest (IHCA); bag-valve-mask (BVM); tidal volume; ventilation rate; intra-arrest ventilation; cardiopulmonary ventilation (CPR); resuscitation; adult
MeSH Terms: conditions — Heart Arrest; Respiratory Aspiration | interventions — Respiration, Artificial; Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: Adult patients (≥18 years) with in-hospital cardiac arrest receiving cardiopulmonary resuscitation.
  Groups will be defined based on observed distribution of ventilation parameters (ventilation rate, tidal volume and minute ventilation).
  Interventions: Other: Positive pressure ventilation during cardiopulmonary resuscitation

INTERVENTIONS:
Other: Positive pressure ventilation during cardiopulmonary resuscitation — The primary exposures of interest are the observed ventilation rate, tidal volume and minute ventilation during cardiopulmonary resuscitation.
  Ventilation data are obtained by inspiratory and expiratory air flow measurements using the EOlife (Archeon, Besançon, France) to which healthcare providers are blinded.
  Other Names: manual ventilation; artificial ventilation; intra-arrest ventilation; bag-valve-mask ventilation; invasive ventilation

SUMMARY:
The goal of this prospective observational study is to learn how ventilation quality parameters during cardiopulmonary resuscitation (CPR) are associated with short-term survival following in-hospital cardiac arrest of adult patients.

The main questions it aims to answer are:

What ventilation volume during CPR is associated with the highest chance of return of spontaneous circulation (ROSC)? What ventilation rate during CPR is associated with the highest chance of ROSC?

Researchers will compare different levels of ventilation rates and volumes that are blindly measured during CPR to see how the observed rates and volumes are associated with survival outcomes and complications.

ELIGIBILITY:
Inclusion Criteria:

1. In-hospital cardiac arrest
2. Age ≥ 18 years
3. >1minute of recorded ventilation data

Exclusion Criteria:

1. Documented do-not-attempt cardiopulmonary resuscitation order
2. Invasive mechanical circulatory support at the time of the cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving ventilation with a bag-valve-mask (BVM) or advanced airway during cardiopulmonary resuscitation for in-hospital cardiac arrest.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Fraction of patients with return of spontaneous circulation (ROSC) | ROSC is assessed immediately following cardiopulmonary resuscitation.
  ROSC is defined as sustained spontaneous circulation with no need for chest compressions for at least 20 minutes.

SECONDARY OUTCOMES:
Fraction of patients surviving until day 30 | Assessed at day 30 after cardiac arrest.
  Patient survival for at least 30 days following cardiac arrest.

OTHER OUTCOMES:
Fraction of patients with pulmonary complications | From date of ROSC until date of intensive care unit discharge or date of death from any cause, whichever came first, assessed up to 30 days.
  Composite endpoint of pulmonary complications after return of spontaneous circulation (ROSC) including acute respiratory distress syndrome (ARDS), aspiration, pneumothorax and hemothorax.
Number of days alive without mechanical ventilation | From date of ROSC until day 30 or date of death from any cause, whichever came first.
  Days patients are alive without receiving mechanical ventilation after return of spontaneous circulation (ROSC).
Number of days alive outside the intensive care unit | From date of ROSC until day 90 or date of death from any cause, whichever came first.
  Days patients are alive outside of the intensive care unit after return of spontaneous circulation (ROSC).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Wittig, MD, Principal Investigator — Department of Clinical Medicine, Aarhus University, Denmark; Department of Medicine, Randers Regional Hospital, Randers, Denmark; Research Center for Emergency Medicine, Aarhus University Hospital, Denmark; Kasper G Lauridsen, MD, PhD, Principal Investigator — Department of Clinical Medicine, Aarhus University, Denmark; Department of Medicine, Randers Regional Hospital, Randers, Denmark; Research Center for Emergency Medicine, Aarhus University Hospital, Denmark;
Locations (11):
- Denmark (10):
  - Hospital of Southern Jutland - Aabenraa, Aabenraa
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Hospital of Southwest Jutland - Esbjerg, Esbjerg
  - Gødstrup Hospital, Gødstrup
  - North Denmark Region Hospital - Hjørring, Hjørring
  - Horsens Regional Hospital, Horsens
  - Odense University Hospital, Odense
  - Randers Regional Hospital, Randers
  - Viborg Regional Hospital, Viborg
- St. Olavs Hospital, Trondheim University Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
The investigators are not permitted to share IPD.